CLINICAL TRIAL: NCT00475761
Title: Breast Radiology Evaluation and Study of Tissues (Breast) Stamp Project
Brief Title: Breast Mammogram and Tissue Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907150; 07-C-N150
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Breast Neoplasms
Keywords: Breast biopsy; Breast imaging; Breast Cancer; Mammographic Density; Natural History
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cohort: Primary clinical- patients referred to diagnostic breast biopsy

SUMMARY:
Background:

Women whose mammograms show a lot of dense areas are more likely to develop breast cancer and to have cancers that are missed by mammograms.

It is unclear why some factors lead to having dense breasts and why having dense breasts increases the risk of developing breast cancer.

Objectives:

To determine why some women s breasts look dense on mammograms.

To determine what types of cells and tissues make up dense areas of breasts and why these tissues may be more likely to become cancerous.

Eligibility:

Women between 40 and 65 years of age who have not had breast cancer or received medicines or radiation for any type of cancer and who are scheduled to undergo a breast biopsy.

Design:

This study is conducted at the University of Vermont, in collaboration with the NCI.

Participants undergo the following:

* Review of their medical records collected over the last 2 years by the Vermont Mammography Registry.
* Participation in a short telephone interview.
* Height and weight measurement.
* Testing of biopsy tissue collected for diagnosis or treatment.
* Future contacts regarding health status for up to 10 years, including review of additional mammograms, removed tissues, questionnaires and medical records collected by the Vermont Mammography Registry during the 10-year study.

Participants may also undergo the following optional procedures:

* Provide a mouthwash sample for genetic testing.
* Provide a blood sample to test for markers of dense mammograms or breast cancer.

DETAILED DESCRIPTION:
High breast density and aging are the strongest risk factors for sporadic breast cancer among women. Although glandular epithelium contributes to mammographic density, non-epithelial tissue components represent its major determinants: adipose tissue is radiolucent and fibrous tissue is dense. The hypothesis is that epidemiologic factors associated with elevated breast density alter the breast microenvironment (ME) (defined as all cells and structures surrounding luminal glandular cells including: myoepithelial cells; basement membrane, stromal fibroblast and myofibroblasts; endothelial cells and pericytes; inflammatory cells, collagens, matrix proteins, growth factors, hormones, and other biochemical components) in a manner that enhances dysregulated proliferation of breast epithelium and ultimately cancer. Specifically, the Investigators propose that epidemiologic factors that lead to increased exposure to hormones and inflammatory mediators alter the ME, leading to both increased breast density and cancer. The critical importance of the ME in carcinogenesis is supported by experimental and clinical data showing that epithelial abnormalities alone are generally insufficient for cancer development without concurrent changes in the ME. The primary aim of this pilot study is to demonstrate the feasibility of collecting the data needed to elucidate the biologic mechanisms that mediate the substantial breast cancer risk associated with high mammographic density. Specifically, the Investigators will develop, fine tune, and validate a complex cross-sectional study protocol to collect risk factor data and biological specimens (blood, buccal cells, tissue fluids, and tissue) required to discover mechanisms and biomarkers that link high mammographic density (as measured quantitatively using computerized methods) to breast cancer risk. They will enroll 250 women between the ages of 40 to 65 years undergoing a radiologically guided biopsy at the University of Vermont, the largest center within the Vermont Breast Cancer Surveillance System (VBCSS), to participate in this pilot study of mammographic density.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for participation in the study are women, ages 40-65 years of age, who are undergoing a radiologically-guided biopsy (stereotactic- ultrasound-guided). We will NOT exclude subjects for current or past use of exogenous hormones; prior hysterectomy or salpingoophorectomy or presentation with a breast mass. Although most biopsies are prompted by a radiologic finding (typically abnormal calcifications or masses), some biopsies are performed for symptoms that are unassociated with a radiologic finding, such as nipple discharge, palpable mass, discomfort, etc. Elevated density per se is not a biopsy indication. ALL women referred for radiologically guided biopsy, irrespective of the indication, will be considered eligible for the pilot study.

EXCLUSION CRITERIA:

We will EXCLUDE women who have a prior history of breast cancer, have had an EXCISIONAL breast biopsy within one year, women who have implants in place, women taking tamoxifen or raloxifene for chemoprevention and women who have received non-surgical treatments for cancers of other organs.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical- patients referred to diagnostic breast biopsy due to an abnormal breast imaging exam.
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2007-05-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of collecting data needed | Dec. 2022
  Feasibility of collecting data needed from pilot to report the preliminary results from the pilot data in published manuscripts.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] Gierach GL, Patel DA, Pfeiffer RM, Figueroa JD, Linville L, Papathomas D, Johnson JM, Chicoine RE, Herschorn SD, Shepherd JA, Wang J, Malkov S, Vacek PM, Weaver DL, Fan B, Mahmoudzadeh AP, Palakal M, Xiang J, Oh H, Horne HN, Sprague BL, Hewitt SM, Brinton LA, Sherman ME. Relationship of Terminal Duct Lobular Unit Involution of the Breast with Area and Volume Mammographic Densities. Cancer Prev Res (Phila). 2016 Feb;9(2):149-58. doi: 10.1158/1940-6207.CAPR-15-0282. Epub 2015 Dec 8. PMID 26645278
- [Background] Gierach GL, Geller BM, Shepherd JA, Patel DA, Vacek PM, Weaver DL, Chicoine RE, Pfeiffer RM, Fan B, Mahmoudzadeh AP, Wang J, Johnson JM, Herschorn SD, Brinton LA, Sherman ME. Comparison of mammographic density assessed as volumes and areas among women undergoing diagnostic image-guided breast biopsy. Cancer Epidemiol Biomarkers Prev. 2014 Nov;23(11):2338-48. doi: 10.1158/1055-9965.EPI-14-0257. Epub 2014 Aug 19. PMID 25139935
- [Background] Horne HN, Sherman ME, Pfeiffer RM, Figueroa JD, Khodr ZG, Falk RT, Pollak M, Patel DA, Palakal MM, Linville L, Papathomas D, Geller B, Vacek PM, Weaver DL, Chicoine R, Shepherd J, Mahmoudzadeh AP, Wang J, Fan B, Malkov S, Herschorn S, Hewitt SM, Brinton LA, Gierach GL. Circulating insulin-like growth factor-I, insulin-like growth factor binding protein-3 and terminal duct lobular unit involution of the breast: a cross-sectional study of women with benign breast disease. Breast Cancer Res. 2016 Feb 18;18(1):24. doi: 10.1186/s13058-016-0678-4. PMID 26893016